CLINICAL TRIAL: NCT03190967
Title: Phase I/II Study of T-DM1 Alone Versus T-DM1 and Metronomic Temozolomide in Secondary Prevention of HER2-Positive Breast Cancer Brain Metastases Following Stereotactic Radiosurgery
Brief Title: T-DM1 Alone Versus T-DM1 and Metronomic Temozolomide in Secondary Prevention of HER2-Positive Breast Cancer Brain Metastases Following Stereotactic Radiosurgery
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The phase II portion was never started as we could no longer get the drug from the manufacturer.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Stanley Lipkowitz, MD, PhD, Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 170115; 17-C-0115
Record Dates: First submitted 2017-06-16; First posted 2017-06-19 (Actual); Results first posted 2023-10-11 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-09

CONDITIONS: Breast Cancer; Brain Metastasis; Brain Cancer
Keywords: Ado-trastuzumab Emtansine; Systemic Control of Disease; Maximum Tolerated Dose; Preventing the Formation of a Metastasis
MeSH Terms: conditions — Breast Neoplasms; Brain Neoplasms | interventions — Ado-Trastuzumab Emtansine; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- 1/Phase I: Ado-trastuzumab (T-DMI) + Temozolomide (TMZ) Dose Escalation (Experimental): T-DM1 + TMZ in dose escalation
  Interventions: Drug: T-DM1; Drug: TMZ
- 2A /Phase II: Arm A, Ado-trastuzumab (T-DMI) Alone (Active Comparator): T-DM1
  Interventions: Drug: T-DM1
- 2B/Phase II /Arm B, Ado-trastuzumab (T-DMI) + Temozolomide (TMZ) (Experimental): T-DM1 + TMZ at recommended phase 2 dose (RP2D)
  Interventions: Drug: T-DM1; Drug: TMZ

INTERVENTIONS:
Drug: T-DM1 — T-DM1 3.6 mg/kg intravenous (IV) every 21 days
  Other Names: Ado-trastuzumab
Drug: TMZ — Phase I: TMZ 30, 40 or 50 mg/m^2 daily Phase II: TMZ at recommended phase 2 dose (RP2D) estimated in Phase I dose escalation part of the study.
  Other Names: Temozolomide
  Arms: 1/Phase I: Ado-trastuzumab (T-DMI) + Temozolomide (TMZ) Dose Escalation; 2B/Phase II /Arm B, Ado-trastuzumab (T-DMI) + Temozolomide (TMZ)

SUMMARY:
Background:

Sometimes breast cancer spreads (metastasizes) to the brain. Researchers want to study new treatments for brain metastases. The drug Temozolomide is approved to treat brain tumors. Researchers want to see if combining it with the drug trastuzumab emtansine (T-DMI) prevents the formation of new metastases in the brain.

Objective:

To study if Temozolomide with T-DM1 lowers the chance of having new metastases in the brain.

Eligibility:

Adults at least 18 years old with a human epidermal growth factor receptor 2 (HER2)-positive breast cancer that has spread to the brain and was recently treated with stereotactic radiation or surgery.

Design:

Participants will be screened with

* Medical history
* Physical exam
* Heart tests
* A scan (computed tomography (CT) that makes a picture of the body using a small amount of radiation
* A scan (magnetic resonance imaging (MRI) that uses a magnetic field to make an image of the brain
* Blood tests.
* Pregnancy test.

The study will be done in 3-week cycles.

All participants will get T-DM1 on Day 1 of every cycle through a small plastic tube inserted in an arm vein.

Some participants will also take Temozolomide capsules by mouth every day.

Participants will keep a medication diary.

During the study, participants will also:

* Repeat most of the screening tests.
* Answer questions about their general well-being and functioning.

Participants will have lumbar puncture at least 2 times. A needle is inserted into the spinal canal low in the back and cerebrospinal fluid is collected. This will be done with local anesthesia and with the help of images.

Participants will be asked to provide tumor samples when available.

Participants will have a follow-up visit about 1 month after stopping the study drug. They will be contacted by telephone or email every 3 months after that.

DETAILED DESCRIPTION:
Background:

* Breast cancer is the most common cancer in women. In the human epidermal growth factor receptor 2 (HER2+) subtype, brain metastases can occur in up to 25-40% of patients.
* The standard therapy for brain metastases continues to be surgery or stereotactic radiosurgery (SRS) and/or whole brain radiation therapy (WBRT).
* Currently, independently of localized or systemic treatment modality, once brain metastases are established, options for treatment are limited, and the disease almost invariably progresses, limiting not only survival but also quality of life in most patients.
* Preclinical literature suggests the hypothesis that preventing the formation of a metastasis by a drug may be more efficacious than attempting to shrink an established lesion.
* Our group has shown in vitro and in vivo in animal models injected with a brain tropic O6-methylguanine DNA methyltransferase (MGMT) + cell line, that even in very low doses temozolomide (TMZ) administered in a prophylactic, metronomic fashion can significantly prevent development of brain metastases.
* We propose a secondary-prevention clinical trial with oral TMZ given to HER2+ breast cancer patients with brain metastases after recent local treatment (SRS or surgical resection) in combination with the anti-HER2 agent T-DM1 for systemic control of disease.

Objectives:

* Phase I (run in): to identify the maximum tolerated dose (MTD) of TMZ when used in combination with T-DM1.
* Phase II: to determine if the combination regimen of trastuzumab emtansine (T-DM1) and temozolomide improves the freedom from distant new brain metastases following stereotactic radiosurgery or surgical resection in HER2-positive breast cancer brain metastases, as compared to T-DM1 alone guided by one-year results as an important benchmark for measuring improvement.

Eligibility:

Phase I:

* Histologically confirmed HER2+ breast cancer.
* Eastern Cooperative Oncology (ECOG) performance status 0-2 and adequate organ and marrow function.
* Brain metastases, treated within 12 weeks of study entry with SRS, resection or WBRT.
* Patients with leptomeningeal metastatic disease are ineligible.
* Patients that are unable to complete a brain MRI with contrast are ineligible.
* Patients with breast tissue expanders must have those removed before enrollment.
* Hepatitis B virus (HBV), hepatitis C virus (HCV) or human immunodeficiency virus (HIV)-positive patients are ineligible.
* Patient with impaired cardiac function or clinically significant cardiac disease are ineligible.
* Corticosteroids will be allowed at enrollment and during the first month of treatment with T-DM1 after SRS, up to a dose of no more than 10mg of dexamethasone daily or equivalent. Patients that need to continue corticosteroids after the initial month will not be allowed to increase the dose after that period and will be taken off protocol.

Phase II:

* Histologically confirmed HER2+ breast cancer.
* ECOG performance status 0-2 and adequate organ and marrow function.
* 1-10 brain metastases, by contrast MRI, treated within 12 weeks of study entry with SRS and/or resection.
* Patients with leptomeningeal metastatic disease are ineligible.
* Patients with history of WBRT are ineligible.
* Patients that are unable to complete a brain MRI with contrast are ineligible.
* Patients with breast tissue expanders must have those removed before enrollment.
* HBV, HCV or HIV-positive patients are ineligible.
* Patient with impaired cardiac function or clinically significant cardiac disease are ineligible.
* Corticosteroids will be allowed at enrollment and during the first month of treatment with T-DM1 after SRS, up to a dose of no more than 10mg of dexamethasone daily or equivalent. Patients that need to continue corticosteroids after the initial month will not be allowed to increase the dose after that period and will be taken off protocol.

Design:

* This is a Phase I/II open label study that will evaluate the potential benefit of TMZ in prevention of new brain metastases in patients with limited brain metastases from HER2+ breast cancer, previously treated with SRS or surgical resection of brain metastases.
* All patients will receive the standard second-line therapy for HER2+ metastatic breast cancer: T-DM1. During phase II patients will be randomized between T-DM1 plus TMZ versus T-DM1 alone.
* Phase I run in: T-DM1 3.6 mg/kg intravenous (IV) every 21 days plus TMZ 30, 40 or 50 mg/m^2 daily.
* Phase II: T-DM1 3.6 mg/kg versus T-DM1 3.6mg/kg plus TMZ at recommended phase 2 dose (RP2D).
* Phase I will follow a standard 3+3 design. Thus, with 3 dose levels, up to 18 patients may be included in the initial safety evaluation.
* In the phase II portion of the trial, a total of 49 evaluable subjects per arm (98 total) will need to be randomized over a 3-year period and followed for an additional 2 years from the date of entry of the last patient, with occurrence of 79 total relapses in both arms combined, in order to have 80% power to compare the curves.

ELIGIBILITY:
* INCLUSION CRITERIA:

Phase 1 Inclusion Criteria

* Patients must have histologically confirmed human epidermal growth factor receptor 2 (HER2)-positive breast cancer for which standard curative measures do not exist or are no longer effective. HER2 testing must have been performed in a laboratory accredited by the College of American Pathologists (CAP) or another accrediting entity.
* Patients must have brain metastases, treated within 12 weeks of study entry with stereotactic radiosurgery (SRS), resection or whole brain radiation therapy (WBRT). A minimum interval of 3 weeks between completion of brain SRS and/or resection and 6 weeks for WBRT and the start of treatment in this trial will be observed to allow proper healing. The presence of concomitant extracranial metastatic disease is allowed for enrollment.
* Corticosteroids will be allowed at enrollment and during the first month of treatment with trastuzumab emtansine (T-DM1) after SRS, up to a dose of no more than 10mg of dexamethasone daily or equivalent. Patients that need to continue corticosteroids after the initial month will be allowed to continue in the protocol treatment if no further increase in dose is necessary. Patients that need increase in dose of corticosteroid after initial month will be taken off protocol treatment.
* Age greater than or equal to18 years. Because breast cancer is not commonly found in pediatric population and no dosing or adverse event data are currently available on the use of temozolomide in combination with T-DM1 in patients <18 years of age, children are excluded from this study, but will be eligible for future pediatric trials.
* Eastern Cooperative Oncology (ECOG) performance status less than or equal to 2 (Karnofsky greater than or equal to 60%, see Appendix A)
* Patients must have normal organ and marrow function as defined below:

  * leukocytes greater than or equal to 3,000/mcL
  * absolute neutrophil count greater than or equal to 1,000/mcL
  * platelets greater than or equal to 100,000/mcL
  * total bilirubin within normal institutional limits
  * Aspartate aminotransferase (AST) serum glutamic-oxaloacetic transaminase (SGOT)/alanine aminotransferase (ALT) serum glutamate pyruvate transaminase (SGPT) <3.0 X institutional upper limit of normal
  * creatinine up to 1.5 upper institutional limits, OR
  * creatinine clearance greater than or equal to 60 mL/min/1.73 m(2) for patients with creatinine levels above institutional normal.
* Alkylating agents as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation and for 7 months (women) or 4 months (men) after treatment completion. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Ability of subject to understand and the willingness to sign a written informed consent document.

Phase 2 Inclusion Criteria

* Patients must have histologically confirmed HER2-positive breast cancer for which standard curative measures do not exist or are no longer effective. HER2 testing must have been performed in a laboratory accredited by the College of American Pathologists (CAP) or another accrediting entity.
* Patients must have 1-10 brain metastases, by contrast magnetic resonance imaging (MRI), treated within 12 weeks of study entry with SRS and/or resection. A minimum interval of 3 weeks between completion of brain SRS and/or resection and the start of treatment in this trial will be observed to allow proper healing. The presence of concomitant extracranial metastatic disease is allowed for enrollment.
* Corticosteroids will be allowed at enrollment and during the first month of treatment with T-DM1 after SRS, up to a dose of no more than 10mg of dexamethasone daily or equivalent. Patients that need to continue corticosteroids after the initial month will be allowed to continue in the protocol treatment if no further increase in dose is necessary. Patients that need increase in dose of corticosteroid after initial month will be taken off protocol treatment.
* Age greater than or equal to 18 years. Because breast cancer is not commonly found in pediatric population and no dosing or adverse event data are currently available on the use of temozolomide in combination with T-DM1 in patients <18 years of age, children are excluded from this study, but will be eligible for future pediatric trials.
* ECOG performance status less than or equal to 2 (Karnofsky greater than or equal to 60%)
* Patients must have normal organ and marrow function as defined below:

  * leukocytes greater than or equal to 3,000/mcL
  * absolute neutrophil count greater than or equal to 1,000/mcL
  * platelets greater than or equal to 100,000/mcL
  * total bilirubin within normal institutional limits
  * AST(SGOT)/ALT(SGPT) <3.0 X institutional upper limit of normal
  * creatinine up to 1.5 upper institutional limits, OR
  * creatinine clearance greater than or equal to 60 mL/min/1.73 m(2) for patients with creatinine levels above institutional normal.
* Alkylating agents as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation and for 7 months (women) or 4 months (men) after treatment completion. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Ability of subject to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

Phase 1 Exclusion Criteria

* Patients who are receiving any other investigational agents.
* Patients unable to speak or understand English, since they cannot complete neurocognitive evaluation.
* Patients with known leptomeningeal metastatic disease.
* Patients with major symptoms or impairments related to brain metastases, such as aphasia or severe confusion, will be excluded per principal investigator (PI) discretion when those symptoms preclude proper neurocognitive evaluation during the study treatment.
* Patients who have received previous treatment with T-DM1 and had systemic progression of disease while on it, are ineligible. Patients receiving treatment with T- DM1 whose only site of disease progression was brain are allowed to enroll in this trial.
* Patients who have received chemotherapy in the previous 3 weeks (6 weeks for nitrosoureas or mitomycin).
* Hepatitis B virus (HBV), Hepatitis B surface antigen positive (HBs Ag positive) or hepatitis C virus (HCV) (anti-HCV positive) patients are ineligible because of potential reactivation of hepatitis virus with temozolomide use.
* Grade greater than or equal to 3 peripheral neuropathy according to (National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
* Cerebral Vascular Accident (CVA) or Transitory Ischemic Attack (TIA) in the year before enrollment, or presence of residual symptoms from CVA that happened more than a year before.
* Pulmonary Embolism (PE) in the 3 months before enrollment. Anticoagulation is permitted.
* Impaired cardiac function or clinically significant cardiac disease including the following:

  * New York Heart Association grade III or IV congestive heart failure.
  * Myocardial infarction within the last 12 months.
* Subjects with impaired left ventricular ejection fraction (LVEF) (<50%).
* Patients with inability to complete brain MRI studies with contrast.
* Patients with breast tissue expanders must have those removed before enrollment.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to temozolomide or T-DM1. Patients who are tolerating TDM1 successfully with pre-medications and slower infusion will be allowed.
* Patients receiving medications that are strong cytochrome P450 3A4 (CYP3A4) inhibitors or inducers are ineligible. In vitro studies indicate that DM1, the cytotoxic component of T-DM1, is metabolized mainly by CYP3A4 and to a lesser extent by cytochrome P450 3A5 (CYP3A5). Concomitant use of strong CYP3A4 inhibitors with T-DM1 should be avoided due to the potential for an increase in DM1 exposure and toxicity. Consider an alternate medication with no or minimal potential to inhibit CYP3A4. Lists including medications and substances known or with the potential to interact with CYP3A4 isoenzymes are provided in Appendix B.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, that would limit compliance with study requirements.
* Pregnant women are excluded from this study because temozolomide is an alkylating agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with temozolomide and/or T-DM1, breastfeeding should be discontinued if the mother is treated with either of those agents. These potential risks may also apply to other agents used in this study.
* human immunodeficiency virus (HIV)-positive patients are excluded because these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy.
* Patients with any other concomitant invasive malignancies are ineligible. Prior invasive cancers treated with curative intent, and with no evidence of recurrent disease, may be eligible after principal investigator (PI) evaluation. Patients with treated limited stage basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the breast or cervix are eligible.

Phase 2 Exclusion Criteria

* Patients who are receiving any other investigational agents.
* Patients unable to speak or understand English, since they cannot complete neurocognitive evaluation.
* Patients with known leptomeningeal metastatic disease.
* Patients previously treated with whole brain radiation therapy (WBRT).
* Patients with major symptoms or impairments related to brain metastases, such as aphasia or severe confusion, will be excluded per PI discretion when those symptoms preclude proper neurocognitive evaluation during the study treatment.
* Patients who have received previous treatment with T-DM1 and had systemic progression of disease while on it, are ineligible. Patients receiving treatment with T- DM1 whose only site of disease progression was brain are allowed to enroll in this trial.
* Patients who have received chemotherapy in the previous 3 weeks (6 weeks for nitrosoureas or mitomycin).
* HBV (HBs Ag positive) or HCV (anti-HCV positive) patients are ineligible because of potential reactivation of hepatitis virus with temozolomide use.
* Grade greater than or equal to 3 peripheral neuropathy according to (NCI CTCAE) version 4.0.
* Cerebral Vascular Accident (CVA) or Transitory Ischemic Attack (TIA) in the year before enrollment, or presence of residual symptoms from CVA that happened more than a year before.
* Pulmonary Embolism (PE) in the 3 months before enrollment. Anticoagulation is permitted.
* Impaired cardiac function or clinically significant cardiac disease including the following:

  * New York Heart Association grade III or IV congestive heart failure.
  * Myocardial infarction within the last 12 months.
  * Subjects with impaired LVEF (<50%).
  * Patients with inability to complete brain MRI studies with contrast.
  * Patients with breast tissue expanders must have those removed before enrollment.
  * History of allergic reactions attributed to compounds of similar chemical or biologic composition to temozolomide or T-DM1. Patients who are tolerating TDM1 successfully with pre-medications and slower infusion will be allowed.
* Patients receiving medications that are strong CYP3A4 inhibitors or inducers are ineligible. In vitro studies indicate that DM1, the cytotoxic component of T-DM1, is metabolized mainly by CYP3A4 and to a lesser extent by CYP3A5. Concomitant use of strong CYP3A4 inhibitors with T-DM1 should be avoided due to the potential for an increase in DM1 exposure and toxicity. Consider an alternate medication with no or minimal potential to inhibit CYP3A4. Lists including medications and substances known or with the potential to interact with CYP3A4 isoenzymes are provided in Appendix B.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, that would limit compliance with study requirements.
* Pregnant women are excluded from this study because temozolomide is an alkylating agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with temozolomide and/or T-DM1, breastfeeding should be discontinued if the mother is treated with either of those agents. These potential risks may also apply to other agents used in this study.
* HIV-positive patients are excluded because these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy.
* Patients with any other concomitant invasive malignancies are ineligible. Prior invasive cancers treated with curative intent, and with no evidence of recurrent disease, may be eligible after PI evaluation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-04-18 (Actual); Primary Completion 2021-06-28 (Actual); Study Completion 2023-06-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanley Lipkowitz, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request. In addition, all large-scale genomic sequencing data will be shared with subscribers to the database of Genotypes and Phenotypes (dbGaP).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data are available during the study and indefinitely. Genomic data are available once genomic data are uploaded per protocol Genomic Data Sharing (GDS) plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to Biomedical Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI). Genomic data are made available via the database of Genotypes and Phenotypes (dbGaP) through requests to the data custodians.

REFERENCES:
- [Background] Swain SM, Kim SB, Cortes J, Ro J, Semiglazov V, Campone M, Ciruelos E, Ferrero JM, Schneeweiss A, Knott A, Clark E, Ross G, Benyunes MC, Baselga J. Pertuzumab, trastuzumab, and docetaxel for HER2-positive metastatic breast cancer (CLEOPATRA study): overall survival results from a randomised, double-blind, placebo-controlled, phase 3 study. Lancet Oncol. 2013 May;14(6):461-71. doi: 10.1016/S1470-2045(13)70130-X. Epub 2013 Apr 18. PMID 23602601
- [Background] Bartsch R, Berghoff AS, Vogl U, Rudas M, Bergen E, Dubsky P, Dieckmann K, Pinker K, Bago-Horvath Z, Galid A, Oehler L, Zielinski CC, Gnant M, Steger GG, Preusser M. Activity of T-DM1 in Her2-positive breast cancer brain metastases. Clin Exp Metastasis. 2015 Oct;32(7):729-37. doi: 10.1007/s10585-015-9740-3. Epub 2015 Aug 25. PMID 26303828
- [Background] Gelmon KA, Boyle FM, Kaufman B, Huntsman DG, Manikhas A, Di Leo A, Martin M, Schwartzberg LS, Lemieux J, Aparicio S, Shepherd LE, Dent S, Ellard SL, Tonkin K, Pritchard KI, Whelan TJ, Nomikos D, Nusch A, Coleman RE, Mukai H, Tjulandin S, Khasanov R, Rizel S, Connor AP, Santillana SL, Chapman JA, Parulekar WR. Lapatinib or Trastuzumab Plus Taxane Therapy for Human Epidermal Growth Factor Receptor 2-Positive Advanced Breast Cancer: Final Results of NCIC CTG MA.31. J Clin Oncol. 2015 May 10;33(14):1574-83. doi: 10.1200/JCO.2014.56.9590. Epub 2015 Mar 16. PMID 25779558
- [Result] Jenkins S, Zhang W, Steinberg SM, Nousome D, Houston N, Wu X, Armstrong TS, Burton E, Smart DD, Shah R, Peer CJ, Mozarsky B, Arisa O, Figg WD, Mendoza TR, Vera E, Brastianos P, Carter S, Gilbert MR, Anders CK, Connolly RM, Tweed C, Smith KL, Khan I, Lipkowitz S, Steeg PS, Zimmer AS. Phase I Study and Cell-Free DNA Analysis of T-DM1 and Metronomic Temozolomide for Secondary Prevention of HER2-Positive Breast Cancer Brain Metastases. Clin Cancer Res. 2023 Apr 14;29(8):1450-1459. doi: 10.1158/1078-0432.CCR-22-0855. PMID 36705597
- [Result] Zimmer AS, Steinberg SM, Smart DD, Gilbert MR, Armstrong TS, Burton E, Houston N, Biassou N, Gril B, Brastianos PK, Carter S, Lyden D, Lipkowitz S, Steeg PS. Temozolomide in secondary prevention of HER2-positive breast cancer brain metastases. Future Oncol. 2020 May;16(14):899-909. doi: 10.2217/fon-2020-0094. Epub 2020 Apr 9. PMID 32270710
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2017-C-0115.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The phase II portion was never started as we could no longer get the drug from the manufacturer.
Groups:
- Level 1 Phase I: Ado-trastuzumab (T-DMI) 3.6 mg/kg + Temozolomide (TMZ) 30 mg/m^2: Level 1: T-DM1 3.6 mg/kg intravenous (IV) every 21 days; Temozolomide 30 mg/m^2 by mouth (PO) daily
- Level 2 Phase I: Ado-trastuzumab (T-DMI) 3.6 mg/kg + Temozolomide (TMZ) 40 mg/m^2: Level 2: T-DM1 3.6 mg/kg intravenous (IV) every 21 days; Temozolomide 40 mg/ m^2 by mouth (PO) daily
- Level 3 Phase I: Ado-trastuzumab (T-DMI) 3.6 mg/kg + Temozolomide (TMZ) 50 mg/m^2: Level 3: T-DM1 3.6 mg/kg intravenous (IV) every 21 days; Temozolomide 50 mg/ m^2 by mouth (PO) daily
- Phase II Arm A: Ado-trastuzumab (T-DMI) Alone: Ado-trastuzumab (T-DMI) Alone
- Phase II Arm B: Ado-trastuzumab (T-DMI) + Temozolomide (TMZ): Ado-trastuzumab (T-DMI) + Temozolomide (TMZ)
Period: Level 1 Dose Escalation
Arm/Group | Level 1 Phase I: Ado-trastuzumab (T-DMI) 3.6 mg/kg + Temozolomide (TMZ) 30 mg/m^2 | Level 2 Phase I: Ado-trastuzumab (T-DMI) 3.6 mg/kg + Temozolomide (TMZ) 40 mg/m^2 | Level 3 Phase I: Ado-trastuzumab (T-DMI) 3.6 mg/kg + Temozolomide (TMZ) 50 mg/m^2 | Phase II Arm A: Ado-trastuzumab (T-DMI) Alone | Phase II Arm B: Ado-trastuzumab (T-DMI) + Temozolomide (TMZ)
Started | 3 | 0 | 0 | 0 | 0
Completed | 3 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Level 2
Arm/Group | Level 1 Phase I: Ado-trastuzumab (T-DMI) 3.6 mg/kg + Temozolomide (TMZ) 30 mg/m^2 | Level 2 Phase I: Ado-trastuzumab (T-DMI) 3.6 mg/kg + Temozolomide (TMZ) 40 mg/m^2 | Level 3 Phase I: Ado-trastuzumab (T-DMI) 3.6 mg/kg + Temozolomide (TMZ) 50 mg/m^2 | Phase II Arm A: Ado-trastuzumab (T-DMI) Alone | Phase II Arm B: Ado-trastuzumab (T-DMI) + Temozolomide (TMZ)
Started | 0 | 3 | 0 | 0 | 0
Completed | 0 | 3 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Level 3
Arm/Group | Level 1 Phase I: Ado-trastuzumab (T-DMI) 3.6 mg/kg + Temozolomide (TMZ) 30 mg/m^2 | Level 2 Phase I: Ado-trastuzumab (T-DMI) 3.6 mg/kg + Temozolomide (TMZ) 40 mg/m^2 | Level 3 Phase I: Ado-trastuzumab (T-DMI) 3.6 mg/kg + Temozolomide (TMZ) 50 mg/m^2 | Phase II Arm A: Ado-trastuzumab (T-DMI) Alone | Phase II Arm B: Ado-trastuzumab (T-DMI) + Temozolomide (TMZ)
Started | 0 | 0 | 6 | 0 | 0
Completed | 0 | 0 | 6 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Level 1 Phase I: Ado-trastuzumab (T-DMI) 3.6 mg/kg + Temozolomide (TMZ) 30 mg/m^2 | Level 2 Phase I: Ado-trastuzumab (T-DMI) 3.6 mg/kg + Temozolomide (TMZ) 40 mg/m^2 | Level 3 Phase I: Ado-trastuzumab (T-DMI) 3.6 mg/kg + Temozolomide (TMZ) 50 mg/m^2 | Total
Number analyzed (Participants) | 3 | 3 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 6 | 9
  >=65 years | 2 | 1 | 0 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.11 (3.93) | 61.19 (7.54) | 51.78 (5.47) | 56.47 (7.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6 | 12
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 2 | 5 | 10
  Unknown or Not Reported | 0 | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 0 | 2
  White | 2 | 1 | 6 | 9
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Phase I: Maximum Tolerated Dose (MTD) of Temozolomide (TMZ) When Used With T-DM1 (Ado-trastuzumab)
Description: Maximum tolerated dose of TMZ when used in combination with T-DM1. MTD is defined as the dose level at which 0 or 1 participant in 6 has a dose limiting toxicity (DLT). A DLT is defined as grade 3 or higher non-hematologic adverse events excluding grade 3 hypertension controlled with anti-hypertensive therapy; or grade 3 asymptomatic electrolytes imbalance; grade 3 endocrinopathy; grade 3 asymptomatic increase in aspartate aminotransferase or alanine aminotransferase; and transient (lasting less than <48 hours) nausea, emesis, or diarrhea if corrected with conservative measures within 24-48 hours. A hematologic grade 4 neutropenia of ≥ 7 days duration, grade ≥ 3 thrombocytopenia, and all other grade 4 hematologic toxicities excluding grade 4 lymphopenia, or leukopenia in the absence of grade 3 or higher neutropenia. Grade 3 is severe. Grade 4 is life-threatening.
Time Frame: first 21 days of treatment
Measure: Number; unit: mg/m^2
Groups:
- All Participants: All participants who received at least one dose of Temozolomide at 30, 40 or 50 mg/m^2 by mouth (PO) daily.
Arm/Group | All Participants
Number analyzed (Participants) | 12
mg/m^2 | 40

2. Primary Outcome: Phase II: Median Amount of Time Participant Survives Without New Brain Lesions After Starting Treatment
Description: Median time to progression. Progression was assessed using the Response Assessment in Neuro-oncology Brain Metastases (RANO-BM) Criteria for evaluation of brain lesions, and the Response Evaluation Criteria in Solid Tumors (RECIST) for systemic evaluation. Progression is a 25% increase in the sum of products of all measurable lesions observed over baseline if no decrease. Or appearance of new lesions, or failure to return for evaluation due to death or deteriorating condition.
Time Frame: From the start of treatment until new brain lesions
Population: This outcome measure was not done because the trial was terminated early due to withdrawal of drug support for the planned randomized phase II cohorts. Data was never collected.
Arm/Group | Phase II Arm A: Ado-trastuzumab (T-DMI) Alone | Phase II Arm B: Ado-trastuzumab (T-DMI) + Temozolomide (TMZ)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Phase I: Number of Participants With Grade 3 and/or Grade 4 Adverse Events
Description: Adverse events were assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). Grade 3 is severe. Grade 4 is life-threatening.
Time Frame: Evaluated at the beginning of every cycle while on study, for an average of 9.6 months (range 2.8-33.9 months).
Measure: Count of Participants; unit: Participants
Groups:
- Level 3 Phase I:Ado-trastuzumab (T-DMI) 3.6 mg/kg + Temozolomide (TMZ) 50 mg/m^2: Level 3: T-DM1 3.6 mg/kg intravenous (IV) every 21 days; Temozolomide 50 mg/ m^2 by mouth (PO) daily
Arm/Group | Level 1 Phase I: Ado-trastuzumab (T-DMI) 3.6 mg/kg + Temozolomide (TMZ) 30 mg/m^2 | Level 2 Phase I: Ado-trastuzumab (T-DMI) 3.6 mg/kg + Temozolomide (TMZ) 40 mg/m^2 | Level 3 Phase I:Ado-trastuzumab (T-DMI) 3.6 mg/kg + Temozolomide (TMZ) 50 mg/m^2
Number analyzed (Participants) | 3 | 3 | 6
Participants
  Grade 3 Anemia | 0 | 1 | 0
  Grade 3 Aspartate aminotransferase increased | 0 | 0 | 1
  Grade 3 CD4 lymphocytes decreased | 1 | 1 | 5
  Grade 3 Dysphasia | 1 | 0 | 0
  Grade 3 Hypokalemia | 0 | 0 | 1
  Grade 3 Lymphocyte count decreased | 1 | 2 | 5
  Grade 3 Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Malignant Neoplasm-CML | 0 | 0 | 1
  Grade 3 Neutrophil count decreased | 0 | 0 | 1
  Grade 3 Platelet count decreased | 0 | 0 | 1
  Grade 3 Surgical and medical procedures - Other, Lap Cholecystectomy/Hernia Repair | 0 | 0 | 1
  Grade 3 White blood cell decreased | 0 | 0 | 1
  Grade 4 White blood cell decreased | 0 | 0 | 0
  Grade 4 CD4 lymphocytes decreased | 0 | 0 | 2
  Grade 4 Lymphocyte count decreased | 0 | 0 | 2
  Grade 5 | 0 | 0 | 0

4. Secondary Outcome: Phase I: Number of Participants With Dose Limiting Toxicity (DLTs) at Each Dose Level
Description: Number of participants with DLTs at each dose level 30 days after treatment. A DLT is defined as grade 3 or higher non-hematologic adverse events excluding grade 3 hypertension controlled with anti-hypertensive therapy; or grade 3 asymptomatic electrolytes imbalance; grade 3 endocrinopathy; grade 3 asymptomatic increase in aspartate aminotransferase or alanine aminotransferase; and transient (lasting less than <48 hours) nausea, emesis, or diarrhea if corrected with conservative measures within 24-48 hours. A hematologic grade 4 neutropenia of ≥ 7 days duration, grade ≥ 3 thrombocytopenia, and all other grade 4 hematologic toxicities excluding grade 4 lymphopenia, or leukopenia in the absence of grade 3 or higher neutropenia. Grade 3 is severe. Grade 4 is life-threatening.
Time Frame: After first cycle of treatment, up to 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Level 1 Phase I: Ado-trastuzumab (T-DMI) 3.6 mg/kg + Temozolomide (TMZ) 30 mg/m^2 | Level 2 Phase I: Ado-trastuzumab (T-DMI) 3.6 mg/kg + Temozolomide (TMZ) 40 mg/m^2 | Level 3 Phase I:Ado-trastuzumab (T-DMI) 3.6 mg/kg + Temozolomide (TMZ) 50 mg/m^2
Number analyzed (Participants) | 3 | 3 | 6
Participants | 0 | 0 | 0

5. Secondary Outcome: Phase II: Time to Whole Brain Irradiation
Description: Time to whole brain irradiation compared between the two arms and Kaplan-Meier curves constructed with a two-tailed log-rank test used to compare the arms.
Time Frame: At progression
Population: as for outcome 2
Arm/Group | Phase II Arm A: Ado-trastuzumab (T-DMI) Alone | Phase II Arm B: Ado-trastuzumab (T-DMI) + Temozolomide (TMZ)
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Phase I: Median Survival
Description: Median amount of time participants survives after therapy. Survival compared between the two arms and Kaplan-Meier curves constructed with a two-tailed log-rank test used to compare the arms.
Time Frame: From date of first therapy until death, an average of 40.79 months
Measure: Median (Standard Deviation); unit: Months
Arm/Group | Level 1 Phase I: Ado-trastuzumab (T-DMI) 3.6 mg/kg + Temozolomide (TMZ) 30 mg/m^2 | Level 2 Phase I: Ado-trastuzumab (T-DMI) 3.6 mg/kg + Temozolomide (TMZ) 40 mg/m^2 | Level 3 Phase I: Ado-trastuzumab (T-DMI) 3.6 mg/kg + Temozolomide (TMZ) 50 mg/m^2
Number analyzed (Participants) | 3 | 3 | 6
Months | 37.8 (22.6) | 48.4 (7.5) | 38.5 (9.5)

7. Secondary Outcome: Phase I: Standard Time to Progression (TTP)
Description: TTP is the time between the first day of treatment to the day of disease progression. Progression was assessed using the Response Evaluation Criteria in Solid Tumors (RECIST). Progression is at least a 25% increase in the sum of products of all measurable lesions over smallest sum observed, clear worsening of any evaluable disease, appearance of any new lesion/site, or failure to return for evaluation due to death or deteriorating condition.
Time Frame: From first day of treatment to the day of disease progression, an average of 15 months.
Population: TTP was not reached for 1 participant in dose level 1, and 1 participant in dose level 3.
Measure: Mean (Standard Deviation); unit: Months
Groups:
- Level 2 Phase I:Ado-trastuzumab (T-DMI) 3.6 mg/kg + Temozolomide (TMZ) 40 mg/m^2: Level 2: T-DM1 3.6 mg/kg intravenous (IV) every 21 days; Temozolomide 40 mg/ m^2 by mouth (PO) daily
Arm/Group | Level 1 Phase I: Ado-trastuzumab (T-DMI) 3.6 mg/kg + Temozolomide (TMZ) 30 mg/m^2 | Level 2 Phase I:Ado-trastuzumab (T-DMI) 3.6 mg/kg + Temozolomide (TMZ) 40 mg/m^2 | Level 3 Phase I:Ado-trastuzumab (T-DMI) 3.6 mg/kg + Temozolomide (TMZ) 50 mg/m^2
Number analyzed (Participants) | 2 | 3 | 5
Months | 6.95 (1.06) | 16.26 (13.8) | 17.46 (8.6)

8. Secondary Outcome: Phase II: Median Survival
Description: as for outcome 6
Time Frame: At death
Population: as for outcome 2
Arm/Group | Phase II Arm A: Ado-trastuzumab (T-DMI) Alone | Phase II Arm B: Ado-trastuzumab (T-DMI) + Temozolomide (TMZ)
Number analyzed (Participants) | 0 | 0

9. Other Pre Specified Outcome: Phase I: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0)
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 44 months and 27 days for level 1, 28 months and 10 days for level 2, and 40 months and 8 days for level 3.
Measure: Count of Participants; unit: Participants
Arm/Group | Level 1 Phase I: Ado-trastuzumab (T-DMI) 3.6 mg/kg + Temozolomide (TMZ) 30 mg/m^2 | Level 2 Phase I: Ado-trastuzumab (T-DMI) 3.6 mg/kg + Temozolomide (TMZ) 40 mg/m^2 | Level 3 Phase I: Ado-trastuzumab (T-DMI) 3.6 mg/kg + Temozolomide (TMZ) 50 mg/m^2
Number analyzed (Participants) | 3 | 3 | 6
Participants | 3 | 3 | 6

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 44 months and 27 days for level 1, 28 months and 10 days for level 2, and 40 months and 8 days for level 3.
Arm/Group | Level 1 Phase I: Ado-trastuzumab (T-DMI) 3.6 mg/kg + Temozolomide (TMZ) 30 mg/m^2 | Level 2 Phase I: Ado-trastuzumab (T-DMI) 3.6 mg/kg + Temozolomide (TMZ) 40 mg/m^2 | Level 3 Phase I: Ado-trastuzumab (T-DMI) 3.6 mg/kg + Temozolomide (TMZ) 50 mg/m^2
All-Cause Mortality (participants affected / at risk) | 2/3 | 1/3 | 1/6
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/3 | 1/6
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Level 1 Phase I: Ado-trastuzumab (T-DMI) 3.6 mg/kg + Temozolomide (TMZ) 30 mg/m^2 (N=3) | Level 2 Phase I: Ado-trastuzumab (T-DMI) 3.6 mg/kg + Temozolomide (TMZ) 40 mg/m^2 (N=3) | Level 3 Phase I: Ado-trastuzumab (T-DMI) 3.6 mg/kg + Temozolomide (TMZ) 50 mg/m^2 (N=6)
Dysphasia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Malignant Neoplasm -CML (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Level 1 Phase I: Ado-trastuzumab (T-DMI) 3.6 mg/kg + Temozolomide (TMZ) 30 mg/m^2 (N=3) | Level 2 Phase I: Ado-trastuzumab (T-DMI) 3.6 mg/kg + Temozolomide (TMZ) 40 mg/m^2 (N=3) | Level 3 Phase I: Ado-trastuzumab (T-DMI) 3.6 mg/kg + Temozolomide (TMZ) 50 mg/m^2 (N=6)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 2 (3) | 0 (0) | 1 (2)
Alanine aminotransferase increased (Investigations) | 3 (5) | 1 (6) | 4 (19)
Alkaline phosphatase increased (Investigations) | 3 (7) | 2 (6) | 4 (14)
Allergic reaction (Immune system disorders) | 1 (1) | 1 (2) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (6) | 2 (7) | 3 (15)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 3 (7) | 2 (7) | 5 (16)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2)
Blood bilirubin increased (Investigations) | 1 (2) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
CD4 lymphocytes decreased (Investigations) | 1 (16) | 2 (13) | 5 (26)
Concentration impairment (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2) | 5 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 1 (2) | 1 (3) | 3 (6)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 1 (2) | 2 (4)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dysesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Edema face (General disorders) | 1 (1) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 1 (2) | 1 (2) | 0 (0)
Electrocardiogram QT corrected interval prolonged (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Endocrine disorders - Other, Elevated TSH (Endocrine disorders) | 0 (0) | 1 (2) | 1 (1)
Endocrine disorders - Other, TSH increase only (Endocrine disorders) | 1 (4) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1) | 2 (2)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Eye disorders - Other, Diplopia (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Eye disorders - Other, L eye twitching (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Eye disorders - Other, Red/tenderness. L eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eye disorders - Other, Twitchy Eye-bilateral (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Eye disorders - Other, sunburn to eyes (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (2) | 2 (2) | 3 (5)
Fever (General disorders) | 1 (1) | 0 (0) | 1 (1)
Flu like symptoms (General disorders) | 0 (0) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
GGT increased (Investigations) | 1 (1) | 1 (1) | 4 (9)
Gastrointestinal disorders - Other, Tongue Ulcers (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hallucinations (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (4) | 3 (3)
Hematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatobiliary disorders - Other, Gallbladder Dyskinesia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (3)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 1 (5) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 2 (6) | 0 (0) | 4 (13)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (2) | 1 (1) | 1 (5)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 4 (5)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, Pain, Red, Swollen L toe & nail (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infections and infestations - Other, Shingles (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Infections and infestations - Other, White Blood Ct. Increased (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Injection site reaction (General disorders) | 0 (0) | 1 (1) | 0 (0)
Investigations - Other, specify (Investigations) | 0 (0) | 0 (0) | 1 (1)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Keratitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 1 (2)
Localized edema (General disorders) | 1 (1) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 3 (26) | 3 (29) | 5 (41)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, Leg Cramp/Abd Cramps (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, Leg Cramps (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Nail discoloration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 3 (3)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (2) | 6 (8)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Lump- back, R side (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Neuroma, foot (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, R breast Calcifications (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (20) | 1 (1) | 2 (6)
Otitis externa (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 2 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (2) | 1 (1) | 4 (5)
Platelet count decreased (Investigations) | 2 (3) | 2 (9) | 6 (35)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (2)
Respiratory, thoracic and mediastinal disorders - Other, Cold/Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, Head cold (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Serum amylase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Sinus pain (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Eczema/Seborrheic Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Erythematous Skin rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Ingrown Right nail (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Nodules/spots on dorsal hands (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Rash, Seborrheic Dermatitis, R arm (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Tick Bite (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, red spot from tick bite (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Surgical and medical procedures - Other, Lap Cholecystectomy/Hernia Repair (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (4) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2)
Urinary urgency (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1) | 5 (7)
Watering eyes (Eye disorders) | 1 (3) | 0 (0) | 0 (0)
Weight loss (Investigations) | 1 (3) | 3 (5) | 4 (7)
White blood cell decreased (Investigations) | 2 (26) | 3 (16) | 4 (28)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-06-06): https://cdn.clinicaltrials.gov/large-docs/67/NCT03190967/Prot_SAP_000.pdf
  • Informed Consent Form (2022-07-12): https://cdn.clinicaltrials.gov/large-docs/67/NCT03190967/ICF_001.pdf